CLINICAL TRIAL: NCT07357545
Title: A Randomized, Double-blind and Active-controlled Phase Ⅰ/Ⅲ Clinical Trial to Evaluate Immunogenicity and Safety of Rabies Vaccine (Vero Cell) for Human Use, Freeze-dried, Administered With Different Immunization Schedules in Healthy Individuals Aged 10-60 Years
Brief Title: Immunogenicity and Safety Assessment of Rabies Vaccine (Vero Cell) for Human Use, Freeze-dried
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BA-CT-001; PRO-PVRV-sf-3001
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rabies (Healthy Volunteers)
Keywords: rabies vaccine; serum-free
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sinovac rabies vaccine - 5 doses (Experimental): Subjects will be randomly assigned to receive 5 doses of Sinovac rabies vaccine on Day 0,3,7,14,28
  Interventions: Biological: Sinovac rabies vaccine
- Sinovac rabies vaccine - 4-1 doses (Experimental): Subjects will be randomly assigned to receive 4 doses of Sinovac rabies vaccine on Day 0,3,7,14
  Interventions: Biological: Sinovac rabies vaccine
- Sinovac rabies vaccine - 4-2 doses (Experimental): Subjects will be randomly assigned to receive 4 doses of Sinovac rabies vaccine on Day 0,3,7,28
  Interventions: Biological: Sinovac rabies vaccine
- Marketed rabies vaccine - 5 doses (Active Comparator): Subjects will be randomly assigned to receive 5 doses of a marketed rabies vaccine in China on Day 0,3,7,14,28
  Interventions: Biological: Marketed rabies vaccine

INTERVENTIONS:
Biological: Sinovac rabies vaccine — Rabies Vaccine (Serum-free Vero Cell), Freeze-dried using three types of PEP schedules
  Arms: Sinovac rabies vaccine - 4-1 doses; Sinovac rabies vaccine - 4-2 doses; Sinovac rabies vaccine - 5 doses
Biological: Marketed rabies vaccine — A markted Rabies Vaccine using 5 doses of PEP schedules
  Arms: Marketed rabies vaccine - 5 doses

SUMMARY:
To evaluate the immunogenicity and safety of different post-exposure prophylaxis (PEP) schedules of Sinovac rabies vaccine, in comparison with a marked rabies vaccinein china, in subjects aged 10-60 years old.

DETAILED DESCRIPTION:
This clinical trial is designed as a randomized, blinded, homologous vaccine-controlled and non-inferiority trial, which consists of two parts.

Part 1 (Pilot Study):

First, 20 subjects aged 18-60 years are enrolled to receive the trial vaccine (Sinovac rabies vaccine) according to the 5-dose schedule on Days 0, 3, 7, 14 and 28. A preliminary safety assessment is conducted on Day 7 after the third dose (before the fourth dose). If the incidence of Grade 3 and above AEs does not exceed 15%, and no death or life-threatening SAE related to vaccination occurs, another 20 subjects aged 10-17 years are enrolled. A safety assessment is performed again on Day 7 after full-course vaccination. If the incidence of Grade 3 and above AEs during the entire observation period does not exceed 15%, and no death or life-threatening SAE related to vaccination occurs, the trial proceeds to Part 2. All subjects are observed for safety up to 6 months after full-course vaccination.

Part 2:

A total of 2,000 subjects are enrolled, and randomized at a 1:1:1:1 ratio, 500 in the 5-dose trial group, 500 in the 5-dose control group, 500 in the 4-dose trial group 1, and 500 in the 4-dose trial group 2. The subjects in the 5-dose trial group and the 5-dose control group receive one dose of the trial vaccine or control vaccine (a marketed rabies vaccine in China) on Days 0, 3, 7, 14 and 28, respectively. The subjects in the 4-dose trial group 1 receive one dose of the trial vaccine on Days 0, 3, 7 and 14; and the subjects in the 4-dose test group 2 receive one dose of the trial vaccine on Days 0, 3, 7 and 28.

Blood samples were collected on Day 0, 14, 28, 42, as well as 3 and 6 months after the full-course vaccination, which was for testing serum neutralizing antibodies are detected using the Rapid Fluorescent Focus Inhibition Test (RFFIT). Solicited AEs within 0-7 days after each dose, unsolicited AEs from the first dose to 30 days after full-course vaccination, and all SAEs from the first dose to 6 months after full-course vaccination are collected.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 10-60 years at enrollment;
2. Volunteers and/or their guardians voluntarily agree to participate in the study and sign the ICF.
3. Volunteers and their families can comply with the protocol requirements for study follow-up (no plans for long-term absence or relocation from the study area);
4. Female volunteers are not pregnant or lactating (negative urine pregnancy test before vaccination) and have no pregnancy plan within 2 months after enrollment;
5. Axillary temperature ≤ 37.2°C.

Exclusion Criteria:

1. History of injection with rabies vaccine and specific passive immune preparations, or history of dog or other mammal bites/scratches (Category II exposure or above) within the past year;
2. History of severe allergies requiring medical intervention from previous vaccinations; other severe allergies, such as allergic shock, angioneurotic edema, allergic purpura, local allergic necrotic reaction (Arthus reaction), severe urticaria, and angioneurotic edema;
3. Pyrexia (axillary temperature > 38.5°C) within 3 days before the first dose vaccination; suffering from acute or chronic infectious diseases (active tuberculosis, viral hepatitis) or in the acute exacerbation phase of any chronic disease;
4. Having received blood/blood-related products or immunoglobulins within 3 months before the first dose vaccination; or planning to use such products within 1 month after the last dose vaccination;
5. Having received live attenuated vaccine within 14 days or any vaccine within 7 days before the first dose vaccination;
6. Any condition (e.g., splenectomy) leading to asplenia or functional asplenia;
7. Diagnosed with congenital or acquired immunodeficiency (HIV), or received immunosuppressant therapy within 3 months (e.g., long-term systemic glucocorticoid use ≥ 14 days, dose ≥ 2 mg/kg/day or ≥ 20 mg/day prednisone or equivalent);
8. Severe congenital anomaly, autoimmune disease, genetic disease; severe heart disorder, kidney disease, diabetes, or other severe chronic disease;
9. History of convulsion, epilepsy, or psychotic disorder;
10. Contraindications for intramuscular injection (e.g., diagnosed thrombocytopenia, any coagulopathy, or anticoagulant therapy);
11. Hypertension unable to be controlled with drugs, such as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg during physical examination before enrollment (for adults aged 18 and above);
12. Currently participating in a clinical study of another investigational or unregistered product (drug or vaccine) or planning to participate in other clinical studies before the end of this clinical study;
13. Any condition of the volunteer that may interfere with the assessment of the study purpose as deemed by the investigator.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2040 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of rabies neutralizing antibodies in pre-vaccination negative subjects of each group | Day 14 after the first dose vaccination
Seroconversion rate of serum rabies neutralizing antibody in pre-vaccination negative subjects of each group | Day 42 after the first dose vaccination
GMC of rabies neutralizing antibodies in pre-vaccination negative subjects of each group | Day 14 after the first dose vaccination

SECONDARY OUTCOMES:
GMC of serum rabies neutralizing antibody in pre-vaccination negative subjects of each group | Day 42 after the first dose vaccination
Seroconversion rate of serum rabies neutralizing antibody in pre-vaccination negative subjects of each group | Day 28 after the first dose vaccination.
Seropositive rate of serum rabies neutralizing antibody in Months 3 and 6 post-full-course vaccination for each group | Months 3 and 6 post-full-course vaccination
Incidence of adverse events. | Up to 30 days after the last-dose vaccination for AEs
GMC of serum rabies neutralizing antibody in pre-vaccination negative subjects of each group | Day 28 after the first dose vaccination.
GMC of serum rabies neutralizing antibody in Months 3 and 6 post-full-course vaccination for each group | Months 3 and 6 post-full-course vaccination
Incidence of serious adverse events. | Up to 6 months after the last-dose vaccination for SAEs;

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dazhu County Center for Disease Control and Prevention, Dazhou
  - Yuechi County Center for Disease Control and Prevention, Guang’an

IPD SHARING:
Plan to Share IPD: No